CLINICAL TRIAL: NCT01689506
Title: Prospective Randomised Controlled Open-label Explorative Multi-centre Pilot Trial of Volulyte®-Supplemented Versus Albumin-supplemented Fluid Resuscitation for Major Burns
Brief Title: Fluid Resuscitation in Patients Suffering From Burns Injury
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to low recruitment
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VOLU-011-C P4; 2011-005734-18 (EudraCT Number)
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Hydroxyethyl Starch Derivatives; Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volulyte (Experimental): Volulyte 6%-supplemented arm: 6 % hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution (solution for infusion)
  Interventions: Drug: Volulyte
- Human Serum Albumin (Active Comparator): 5% Albumin-supplemented arm: Human Serum Albumin (HSA 50g/L, solution for infusion)
  Interventions: Drug: Human Serum Albumin

INTERVENTIONS:
Drug: Volulyte — 6 % hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution will be intravenously infused in order to achieve and maintain predefined hemodynamics goals and may be given up to a total daily dose of 50 mL/kg body weight/day.
  Other Names: 6 % hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution
  Arms: Volulyte
Drug: Human Serum Albumin — 5% Human Serum Albumin will be intravenously infused in order to achieve and maintain predefined hemodynamics goals with no daily dose limit.
  Arms: Human Serum Albumin

SUMMARY:
This clinical study compares two fluid resuscitation treatments in patients suffering from burns injury. The treatments are Volulyte® and Human Serum Albumin (HSA) which will be administered as infusion solutions. It will be evaluated whether Volulyte® is effective and safe, and provides any benefit.

DETAILED DESCRIPTION:
Severe burns injury presents a unique resuscitation problem due to simultaneous loss of electrolyte and protein-rich exudate from the burn wound itself and leakage of fluid and protein from the circulation into the interstitial compartment. In the post shock phase of burn resuscitation, patients frequently suffer oedema of unburned tissues and organs and a positive fluid balance of many litres. This pilot study will compare two burns fluid resuscitation regimes (supplementation with 6% HES 130/0.4 in an isotonic electrolyte solution, Volulyte 6%, versus supplementation with Human Serum Albumin, HSA 50g/L) on patient outcome with particular regard to fluid balance at 24 hours after burns injury (primary variable).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age
* 15%≥ Burn Total Body Surface Area Injury ≤60%
* Signed written informed consent from patient or legal representative

Exclusion Criteria:

* Patient age >80 years
* Delay of patient randomisation >8 hours post-burn
* Known pregnancy
* Known renal failure with oliguria or anuria not related to hypovolaemia (e.g. patients receiving dialysis treatment)
* High voltage electrical conduction injury
* Known severe liver disease
* Known fluid overload (hyperhydration), especially in cases of pulmonary oedema and congestive cardiac failure
* Intracranial bleeding (known active or suspicion of intracranial bleeding)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cumulative fluid balance (input-output) | at 24 hours after burns injury

SECONDARY OUTCOMES:
Cumulative fluid balance (input-output) | at 8 hours after burns injury, at 24 hours after randomisation, and until day 7 after burns injury
Oedema monitoring: patient's weight, circumference measurement of unburned limb | once daily until day 7 after burns injury
Urine output | hourly until 24 hours after burns injury, at 24 hours after randomization and, thereafter, once daily until day 7 after burns injury
Haemodynamics | hourly until 24 hours after burns injury, at 24 hours after randomization and, thereafter, 4 times daily until day 7 after burns injury
Bladder pressure | once daily until day 7 after burns injury
Use of vasoactive and inotropic drugs | until 24 hours after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Naiem Moiemen, PhD MD, Principal Investigator — Plastic and Burns Department, University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Queen Elizabeth Medical Centre
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Queen Elizabeth Medical Centre, Birmingham, United Kingdom